CLINICAL TRIAL: NCT02216448
Title: The Benefit of Arthroscopic Simulator Training Versus Operating Room Training in Diagnostic Knee Arthroscopy for Residents With Basic Arthroscopic Skills
Brief Title: Arthroscopy Simulator Training vs OR Training Knee
Acronym: ASTOR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems with simulator
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Dan Prat MD, MD, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SHEBA-14-1236-DP-CTIL
Record Dates: First submitted 2014-07-09; First posted 2014-08-15 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Knee Arthroscopy Skills
Keywords: Arthroscopy skills; Knee; Virtual reality; Simulator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- simulator training (Other): Training knee simulator in Lab
  Interventions: Other: Training knee simulator
- OR training (Other): Training in the OR - 2 knee arthroscopies.
  Interventions: Other: OR Training

INTERVENTIONS:
Other: Training knee simulator — Training in a lab on a virtual reality knee arthroscopy simulator
  Arms: simulator training
Other: OR Training — Training on diagnostic knee arthroscopy in the OR
  Arms: OR training

SUMMARY:
The purpose of this study is to compare between two groups of residents with basic arthroscopic skills in diagnostic knee arthroscopy. The first group will train on a knee arthroscopic simulator in a lab, and the second group will perform diagnostic knee arthroscopy in the operating room. Both groups will be assessed by senior arthroscopy surgeon in the operating room based on selected competencies following the Global Rating System.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic residents

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Global rating scale | completion of training
  About 3 months will be needed for both study arms to complete the training in the arthroscopy lab and in the OR. Then, both will be assessed by the global rating scale for arthroscopy.

SECONDARY OUTCOMES:
simulator parameters | Completion of training
  Secondary outcome measures are technical parameters provided by the simulator for each trainee. At the end of the training sessions, about 3 months from the beginning of the study, this parameters can be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Tel Hashomer, Ramat Gan, Israel